CLINICAL TRIAL: NCT05731232
Title: Effects of Vivatlac Synbiotic in Patients With Irritable Bowel Syndrome - A Randomized, Double-Blind, Placebo-Controlled Clinical Trail
Brief Title: Effects of Vivatlac Synbiotikum in Patients With Irritable Bowel Syndrome
Acronym: ViIBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The President Stanisław Wojciechowski State University of Applied Sciences in Kalisz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Kalisz 2023-02
Record Dates: First submitted 2023-01-31; First posted 2023-02-16 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized allocation to verum or placebo group of similar size
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pacebo (Placebo Comparator): Capsules containing maize starch with identical appearance as verum. One capsule taken per day before bedtime. Treatment duration 12 weeks.
  Interventions: Dietary Supplement: Vivatlac Synbiotikum
- Vivatlac Synbiotikum (Experimental): Vivatlac Synbiotikum for twelve weeks. One capsule containing a mixture of nine different probiotic bacteria with a total amount of 4.5 x 10˄9 colony forming units taken per day before bedtime. Treatment duration 12 weeks.
  Interventions: Dietary Supplement: Vivatlac Synbiotikum

INTERVENTIONS:
Dietary Supplement: Vivatlac Synbiotikum — Each capsule of Vivatlac® Synbiotikum contains a total of 4.5 x 10˄9 colony forming units (CFU) of nine different probiotic bacteria. Probiotic bacteria strains and their CFU amount per capsule are: Lactococcus lactis Ll-23, 9.00 x 10˄8 CFU; Lactobacillus helveticus SP 27, 9.00 x 10˄8 CFU; Bifidobacterium longum Bl-05, 6.75 x 10˄8 CFU; Bifidobacterium breve Bb-03, 4.50 x 10˄8 CFU; Lacticaseibacillus rhamnosus Lr-32, 4.50 x 10˄8 CFU; Streptococcus thermophiles St-21, 4.50 x 10˄8 CFU; Lacticaseibacillus casei Lc-11, 2.25 x 10˄8 CFU; Lactiplantibacillus plantarum Lp-115, 2.25 x 10˄8 CFU; Bifidobacterium bifidum Bb-02, 2.25 x 10˄8 CFU. As a prebiotic component each capsule contains 63 mg of fructooligosaccharides.

SUMMARY:
Multi-centre, randomized, double-blind, placebo-controlled trial investigating the effects of a nine-strain synbiotic (Vivatlac Synbiotikum) in IBS patients.

DETAILED DESCRIPTION:
The study design is a multi-centre, randomized, double-blind, placebo controlled clinical trial in patients diagnosed with IBS. Diagnosis of IBS with the World Gastroenterology Organisation's IBS questionnaire for health care providers. Assessment of severity of IBS by using the IBS Severity of Symptoms Scale (IBS-SSS). IBS patients with moderate to severe IBS will be included into the study (IBS-SSS ≥ 175). A four weeks screening phase is used to evaluate patients' IBS and their capability to report IBS symptoms using a patient diary. The screening phase is followed by treatment with one capsule per day of a nine-strain synbiotic (Vivatlac® Synbiotikum) or placebo for twelve weeks. Each capsule of Vivatlac® Synbiotikum contains a total of 4.5 x 10˄9 colony forming units (CFU) of nine different probiotic bacteria. Probiotic bacteria strains and their CFU amount per capsule are: Lactococcus lactis Ll-23, 9.00 x 10˄8 CFU; Lactobacillus helveticus SP 27, 9.00 x 10˄8 CFU; Bifidobacterium longum Bl-05, 6.75 x 10˄8 CFU; Bifidobacterium breve Bb-03, 4.50 x 10˄8 CFU; Lacticaseibacillus rhamnosus Lr-32, 4.50 x 10˄8 CFU; Streptococcus thermophiles St-21, 4.50 x 10˄8 CFU; Lacticaseibacillus casei Lc-11, 2.25 x 10˄8 CFU; Lactiplantibacillus plantarum Lp-115, 2.25 x 10˄8 CFU; Bifidobacterium bifidum Bb-02, 2.25 x 10˄8 CFU. Effects will be assessed by using the IBS Severity of Symptoms Scale (IBS-SSS), assessment of changes of IBS severity by using the IBS Global Improvement Scale (IBS-GIS) and assessment of IBS relief by using the IBS Adequate Relief scale (IBS-AR) every four weeks. Additional measures will be stool consistency using the Bristol Stool Scale, number of bowel movements, severity of pain, severity of bloating, stool pressure, feeling of incomplete evacuation of stool and adverse events using a patient diary.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed for Irritable Bowel Syndrome using the IBS questionnaire for health care providers of the World Global Gastroenterology Organization
* IBS-SSS ≥ 175 points

Exclusion Criteria:

* patients currently taking products containing probiotics or have taken this kind of products during the last 3 months
* patients currently taking antibiotics or have taken antibiotics during the last 3 months
* patients having a concurrent severe illness (malignancies, uncontrolled hypertension or diabetes, hepatic, renal or cardiac dysfunctions, serious neurological disorders, psychosis, respiratory disorders such as asthma or COPD, hyper- or hypothyroidism
* patients having chronic bowel disorders other than IBS, including inflammatory bowel disease, gastroenteritis, stomach and duodenal cancer, celiac disease
* patient being pregnant or are lactating
* patient being diagnosed to have a lactose intolerance
* patients using motility drugs or dietary fiber supplements withing 2 weeks before study start
* patient taking anti-coagulant medication
* patients have participated in another clinical trial within the last three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Severity of IBS using Severity of Symptoms Scale (IBS-SSS) | Change from baseline after 4, 8 and 12 weeks of treatment
  IBS-Severity Scoring System is a 5-question survey that asks: 1. the severity of abdominal pain, 2. frequency of abdominal pain, 3. severity of abdominal distention, 4.dissatisfaction with bowel habit, and 5. interference with quality of life over the past 10 days. Subjects respond to each question on a 100-point visual analogue scale. Each of the five question generates a maximum score of 100 point, and total scores can range from 0-500 with higher scores indicating severe symptoms. A decrease of 50 points is associated with a clinically meaningful improvement.
Changes of IBS severity using the IBS Global Improvement Scale (IBS-GIS) | Change from baseline after 4, 8 and 12 weeks of treatment
  IBS-Global Improvement Scale asseses changes of IBS symptoms using a patient-defined 7 point Linkert scale ranging from symptoms substantially worse to substantially improved.
  Patients answer the question "Have you felt any change in the severity of your symptoms over the past 7 days compared to how you felt before the medicine was given?
  The answers are recorded based on the 7-point scale:
  * I feel that the symptoms have worsened significantly
  * I feel that the symptoms have moderately worsened
  * I feel that the symptoms have slightly worsened
  * I feel no change
  * I feel a slight improvement
  * I feel moderate improvement
  * I feel significant improvement
  IBS-GIS score indicates: improvement if is >4 or worsening if is<4, no change if is 4
Changes in adequate relief of IBS symptoms (IBS-AR) | Change from baseline after 4, 8 and 12 weeks of treatment
  IBS-Adequate Relief (IBS-AR) is a dichotomous single item that asks participants "Over the past week (7 days) have you had adequate relief of your IBS symptoms? The answer is YES or NO.

SECONDARY OUTCOMES:
Changes in type of stools | Change from baseline weekly for 12 weeks of intervention
  Average consistency of last week's stool assessed weekly before intervention and then weekly duing the treatment period. Type of stools assessed using the Bristol Stool Scale. Bristol Scale is designed to classify faeces into seven groups: type 1-2 indicate constipation, type 3-4 are "normal" stools; type 5-7 indicate diarrhea.
Average number of daily bowel movements during the last week | Change from baseline weekly for 12 weeks of intervention
  Average number of bowel movements per day assessed before intervention and then weekly during the treatment period.
Severity of pain using a five point scale of predefined severity levels | Change from baseline weekly for 12 weeks of intervention
  The severity of pain assessed before intervention and then weekly during the treatment period using a patient-defined 5 point Linkert scale: point 0 - no pain, and 1-4 the severity of pain with higher scores indicating worse pain.
Severity of bloating using a five point scale of predefined severity levels | Change from baseline weekly for 12 weeks of intervention
  The severity of bloating assessed before intervention and then weekly during the treatment period using a patient-defined 5 point Linkert scale: point 0 - no bloating, and points1-4 with higher scores indicating worse bloating.
Stool pressure using a five point scale of predefined severity levels | Change from baseline weekly for 12 weeks of intervention
  The severity of stool pressure assessed before intervention and then weekly during the treatment period using a patient-defined 5 point Linkert scale: point 0 - no stool pressure, and points1-4 with higher scores indicating worse stool pressure.
Feeling of incomplete evacuation of stool | Change from baseline weekly for 12 weeks of intervention
  The feeling of incomplete evacuation of stool assessed before intervention and then weekly during the treatment period using a dichotomous single item that asks participants "Please rate the feeling of incomplete evacuation of stool you have experienced during this week by selecting one of the two answers. Answer are NO SUCH FEELING or THERE IS AN INCOMPLETE BOWEL MOVEMENT.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Piatek, Prof. Dr., Principal Investigator — Calisia University, Kalisz, Poland
Locations (2):
- Poland (2):
  - Family doctor's outpatient clinic "Panacea", Krynki
  - Family doctor's clinic, Stawiszyn

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piatek J, Sommermeyer H, Bernatek M, Ciechelska-Rybarczyk A, Oleskow B, Mikkelsen LS, Barken KB. Persistent infection by Salmonella enterica servovar Typhimurium: are synbiotics a therapeutic option? - a case report. Benef Microbes. 2019 Mar 13;10(2):211-217. doi: 10.3920/BM2018.0080. Epub 2018 Dec 21. PMID 30574800
- [Background] Piatek J, Krauss H, Ciechelska-Rybarczyk A, Bernatek M, Wojtyla-Buciora P, Sommermeyer H. In-Vitro Growth Inhibition of Bacterial Pathogens by Probiotics and a Synbiotic: Product Composition Matters. Int J Environ Res Public Health. 2020 May 11;17(9):3332. doi: 10.3390/ijerph17093332. PMID 32403297
- [Background] Sommermeyer H, Pituch HM, Wultanska D, Wojtyla-Buciora P, Piatek J, Bernatek M. Inhibition of Quinolone- and Multi-Drug-Resistant Clostridioides Difficile Strains by Multi Strain Synbiotics-An Option for Diarrhea Management in Nursing Facilities. Int J Environ Res Public Health. 2021 May 30;18(11):5871. doi: 10.3390/ijerph18115871. PMID 34070727
- [Derived] Sommermeyer H, Chmielowiec K, Bernatek M, Olszewski P, Kopczynski J, Piatek J. Effectiveness of a Balanced Nine-Strain Synbiotic in Primary-Care Irritable Bowel Syndrome Patients-A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Trial. Nutrients. 2024 May 16;16(10):1503. doi: 10.3390/nu16101503. PMID 38794741